CLINICAL TRIAL: NCT00801593
Title: Arthritis of the Temporomandibular Joints in Children With Juvenile Idiopathic Arthritis- Pilot Study on Diagnostic Value of Ultrasonography and Magnetic Resonance Imaging and Influence of Drug Treatment
Brief Title: Magnetic Resonance Imaging Follow-up on Temporomandibular Arthritis in Children With Juvenile Idiopathic Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Nikolay Tzaribachev, Dr., University Children's Hospital, Tuebingen
Other Study IDs: TMJ PROSPECT2008
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2008-12-03 (Estimated); Status verified 2008-12

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: JIA
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with JIA
  Interventions: Procedure: Steroid injection into the TMJs.

INTERVENTIONS:
Procedure: Steroid injection into the TMJs. — In case of otherwise noncontrollable TMJ involvement steroids are injected into arthritic TMJs under MRI guidance.

SUMMARY:
Children with juvenile idiopathic arthritis (JIA) suffer in up to 87% of the cases of arthritis of the temporomandibular joints (TMJs). Magnetic resonance imaging (MRI) is the only modality for the early diagnosis of TMJ involvement.

Aim of the study is to compare symptoms and clinical findings with MRI and ultrasonography results and to describe the action of the current medication on the arthritis of the TMJs.

ELIGIBILITY:
Inclusion Criteria:

* Children with defined JIA.

Exclusion Criteria:

* Children without defined diagnosis of JIA.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with JIA.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
TMJ arthritis on MRI | every three to six months from recruitment to end of study

SECONDARY OUTCOMES:
TMJ arthritis on ultrasound | every three to six months from recruitment to end of study
Action of current medication on TMJ arthritis. | every three to six months from recruitment to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Nikolay Tzaribachev, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Children's Hospital, Tübingen, Baden-Wurttemberg, Germany